CLINICAL TRIAL: NCT01977885
Title: Exercise-Induced Epigenetic Modifications in Obese Aging Women
Acronym: DIVAS2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Georgia (Other)
Responsible Party: Principal Investigator, Ellen Evans, Associate Professor of Kinesiology, University of Georgia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2013106780
Record Dates: First submitted 2013-10-16; First posted 2013-11-07 (Estimated); Last update posted 2015-09-25 (Estimated); Status verified 2015-09

CONDITIONS: Metabolic Syndrome
Keywords: epigenetics; obesity; overweight; high protein diet; exercise; post menopausal women
MeSH Terms: conditions — Metabolic Syndrome; Obesity; Overweight; Motor Activity | interventions — Diet, High-Protein; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- High Protien Diet + Exercise (Experimental): All participants will participate in both interventions (High Protein Diet and Exercise).
  Interventions: Behavioral: High Protein Diet; Behavioral: Exercise

INTERVENTIONS:
Behavioral: High Protein Diet — All participants will be individually counseled by an RD for ~ 4 sessions (30 to 60 minutes)to meet weight loss goals. During the duration of the study, participants will be required to attend a 30 to 60 minute group educational/motivational meeting weekly (first 1 to 2 months) and then biweekly (for the remainder of the study). Diet recommendations will include high quality proteins with an emphasis on lean meats with protein being targeted for every meal and snack. Regarding beef intake specifically, the prescribed diet will include a minimum of one serving of beef per day, which is approximately 3 to 3.5 ounces or ~100 grams. This amount of lean cooked beef provides an average of ~25-30 grams of protein per day (www.beefnutrition.org/leanbeef.aspx). This combined with reducing energy from carbohydrates and fat from other sources will create an overall energy deficit of 500 kcal/day. This diet will also include 5 servings/day of vegetables and 2-3 servings/day of fruit
Behavioral: Exercise — Participants will be prescribed a supervised exercise program with required attendance of 3 nonconsecutive days per week (75 minutes each session). A program that combines flexibility and balance activities, weight bearing endurance exercise (walking) and resistance training to preserve lean mass will be prescribed. With specific regard to strength training, 50% of the resistance work will involve primary muscle groups of the lower body with the main focus being the gluteal and quadriceps groups (squats, lunges, etc.). The remaining 50% of work will dedicate 25% to the core stabilizers with the final 25% being the upper body. Transitions between segments of training will be used for recovery and social support enhancement. Note that all aspects of the exercise intervention will be progressive in intensity (i.e., starting at lower end of intensity or ~50% of maximal capacity), and duration (i.e., from 15 minutes to 35 minutes of exercise and adding a few minutes each session).

SUMMARY:
Our greatest public health challenge is obesity and the co-morbidities of metabolic syndrome (MetS). Age is an established risk factor for MetS and specific to women, data indicates that the prevalence of MetS increases substantially with the menopausal transition with postmenopausal women having a 60% increased risk of MetS. Menopause also contributes to reductions in strength, physical function and often psychological well-being (e.g. fatigue). Obese individuals also have: a) impaired immune function and chronic inflammatory responses associated with changes in the white blood cell population in blood and fat tissues; and, b) increased secretion of and signaling by proteins in their fat cells. Weight loss, which requires an energy deficit through increased physical activity and/or caloric restriction (EX+CR), reduces risk for MetS in older sedentary obese women by reducing insulin resistance and chronic systemic inflammation. Science and clinical practice will be advanced by examining the molecular mechanisms by which EX+CR affects risk for MetS in older women. The primary aim is to determine if CD4+ T cells will report the differential epigenetic reprogramming of relevant gene expression associated with metabolic indices resulting from EX+CR induced weight loss in older women known to be at risk for MetS. This pilot data will be used to generate an NIH proposal of the same topic. A secondary aim is to assess the impact of weight loss on physical function and psychological well-being which will provide pilot data for an additional grant proposal regarding weight management in postmenopausal women.

ELIGIBILITY:
Inclusion Criteria:

1. Volunteer for the study
2. Age between 50 and 64 years
3. Self-identified as White or Caucasian
4. Postmenopausal
5. Sedentary (less than 1 hour each week of planned physical activity and sedentary job)
6. BMI range >/= 25 kg/m2
7. Waist circumference >88cm
8. Weight stable (within 2 kg) for 6 months
9. All allowable medications stable for 3 months
10. Live independently
11. Willing and able to obtain transportation to and from lab sessions
12. Obtains physician clearance to participate in the study

Exclusion Criteria:

1. Tobacco use
2. Normal weight (BMI < 25 kg/m2)
3. Males
4. Dietary restrictions that do not allow for the consumption of beef, as required by our dietary protocol
5. Weight loss surgery and/or weight loss medications usage
6. Mini-mental state exam score < 25
7. Recent or history of unstable CVD
8. Cancer treatment within the last 5 years or active cancer
9. History of lung disease or COPD or severe asthma
10. History or severe arthritis or other medical condition that precludes ability to exercise to level needed by study.
11. Current diagnosis or history of balance disorders
12. History of mental disorders, dementia, clinical depression or other disorders that preclude adherence to protocols.
13. Current weight of 350 pounds or greater, due to weight restrictions on equipment.

Ages: 50 Years to 64 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2013-06; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Change in CD4+T Cells from Baseline to Post-Intervention | Baseline (Week 0), Post-Intervention (Week 24)
  The primary aim is to determine if CD4+ T cells will report the differential epigenetic reprogramming of relevant gene expression associated with metabolic indices resulting from EX+CR induced weight loss in older women known to be at risk for MetS.

SECONDARY OUTCOMES:
Change in Physical Function over 6 Months | Baseline (Week 0), Midpoint (Week 12), Post-Intervention (Week 24)
  A secondary aim is to assess the impact of weight loss on physical function, which will provide pilot data for an additional grant proposal regarding weight management in postmenopausal women.
Change in Psychological Well Being over 6 Months | Baseline (Week 0), Midpoint (Week 12), Post-Intervention (Week 24)
  A battery of psychological assessments will be administered at three time points throughout the study to evaluate possible changes in psychological well being throughout the intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Body Composition and Metabolism Lab, UGA, Ramsey Student Center, Athens, Georgia, United States